CLINICAL TRIAL: NCT05133596
Title: Study of the Evolution of Olfactory Disorders in Patients With Persistent Loss of Smell Following COVID-19
Acronym: ETOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Hopital Lariboisière (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-006; 2021-A02419-32 (Other: ID-RCB)
Record Dates: First submitted 2021-11-23; First posted 2021-11-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease
Keywords: Neuroinflammation; coronavirus; olfaction disorder; evoked potentials
MeSH Terms: conditions — Neuroinflammatory Diseases; Coronavirus Infections; Olfaction Disorders | interventions — Restraint, Physical; Blood Specimen Collection; Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: Adult subjects up to 55 years of age with persistent olfaction disorder after a symptomatic episode of COVID-19.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study population (Experimental): Adult subjects up to 55 years of age with persistent olfaction disorder after a symptomatic episode of COVID-19.
  Interventions: Other: Clinical examination; Other: Blood collection; Other: Olfactory evoked potentials; Other: Brushing of olfactory slits; Other: Neurological examination and neuropsychological assessment; Other: Nasal endoscopy; Other: Assessment of olfactory and taste functions

INTERVENTIONS:
Other: Clinical examination — The investigator will conduct a clinical examination to rule out other causes of olfactory impairment independent of COVID-19. The investigator will also collect the following information: socio-demographic data (age, sex, blood type, weight, height, etc.), history of olfaction disorder symptoms, past or current treatments received and tobacco/alcohol consumption.
Other: Blood collection — 12ml-blood sample
Other: Olfactory evoked potentials — Olfactory evoked potentials will be recorded during olfactory tests.
Other: Brushing of olfactory slits — collection of olfactory slits cells.
Other: Neurological examination and neuropsychological assessment — * MOCA, BREF
  * CVLT
  * WAIS IV, MEM III
  * Right-side and left-side empan, Trail Making Test A and B (TMT), verbal fluency tests, PASAT, Attention Assessment Test
  * Benton's Line Judgement, VOSP
  * Assessment of psychological status, fatigue and screening for psychiatric comorbidities: depression & anxiety scales (HAD scale, mADRS depression scale, STAI anxiety scale), Fatigue Severity Scale.
Other: Nasal endoscopy — Nasal endoscopy
Other: Assessment of olfactory and taste functions — * scales: VAS and TSS
  * Sniffin Stick test

SUMMARY:
The COVID-19 pandemic is a novel medical challenge, particularly because of the systemic nature of this disease. Indeed, COVID-19 affects several organs and systems at once. The brain is affected in several ways: direct infection of nerve cells by SARS-CoV-2, inflammation of the central nervous system, severe systemic inflammation damaging nerve cells, global cerebral ischaemia related to respiratory failure, thromboembolic events related to increased intravascular coagulation and severe psychological stress. As a result, COVID-19 sometimes manifests as neurological and neuropsychiatric symptoms such as dizziness, sleep disturbances, cognitive deficits, delirium, or severe depression.

Sudden loss of smell is a common symptom associated with COVID-19 and SARS-CoV-2 infection of neurons in the olfactory system has been reported in both hamsters and humans. The vast majority of COVID-19 patients recover their olfactory function within a few weeks. However, a significant minority of infected individuals (1 in 5 cases) still suffers from olfactory disorders (anosmia, hyposmia and/or parosmia) several months after the primary infection. These olfactory disorders are frequently associated with depressive behaviour and cognitive complaints. In PET scans, it is even possible to correlate this cognitive dysfunction with hypometabolism of certain brain regions, including the olfactory gyrus.

This project proposes, during one year, to evaluate and follow the evolution of the olfactory capacities of patients suffering from persistent smell disorder since one year (+/- 4 months) following COVID-19. The issue is to study the link between viral persistence in the olfactory sensory organ, chronic inflammation, and central damage to the olfactory system. The follow-up of the evolution of olfactory and neurocognitive capacities, in an integrative way by means of molecular, physiological and behavioural approaches, will inform us on the specificities of "COVID-long" and on the level of peripheral and/or central damage of the olfactory system.

DETAILED DESCRIPTION:
Prospective monocentric descriptive study. Evaluation of COVID-19 patients with persistent loss of smell during 2 visits at 1 year intervals (V1 and V2).

V1 :The following examinations will be carried out specifically for the research.

* Clinical examination;
* Blood sampling;
* Recording of olfactory evoked potentials;
* Neurological examination and neuropsychological assessment;

V2 :

All examinations performed at V1 will be repeated at V2.

If the following examinations are not carried out during care within 3 weeks of V2, they will be carried out as part of the research during this V2 visit.

* Nasal endoscopy ;
* Assessment of olfactory and gustatory functions.

The following explorations will be carried out:

* Passing of two olfactory and gustatory scales; Olfactory and gustatory disorders will be quantified using two scales, the visual analogue scale VAS and the modified TSS;
* Sniffin Stick test.

In addition, MRI data from clinical care will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults < 55 years
* History of symptomatic COVID over 1 year +/- 4 months with a positive PCR diagnosis of SARS-CoV-2
* Olfactory complaint
* Able to understand simple questionnaires in French.
* Subject covered by French Social Security (except for Aide Médicale d'Etat).

Exclusion Criteria:

* Contraindication to nasal swabbing (for morphological reasons, haemostasis disorders, taking aspirin in the 15 days prior to swabbing or anticoagulants, contraindications to the use of a local anaesthetic such as a history of allergy to local anaesthetics or any other reasons judged by the clinical investigator)
* To have been placed in the intensive care unit following COVID-19.
* Known previous nasal-sinus pathology.
* History of psychiatric pathology according to DSM IV criteria, ischaemic, neoplastic, inflammatory, infectious or neurodegenerative (meningitis, encephalopathy, encephalitis, stroke, neurodegenerative disease) known or suspected.
* History of loss of sense of smell prior to COVID infection.
* Patient affiliated to the Aide Médicale d'Etat.
* Person deprived of liberty by judicial or administrative decision, or subject to legal protection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Measurement of olfactory responses by PEO recording and by calculating the TDI score of the Sniffin'stick tests. | 24 months
  To characterise the evolution of the olfactory capacities of patients suffering from persistent odour disorders following SARS-CoV-2 infection over the course of a year.

SECONDARY OUTCOMES:
Measurement of olfactory perception threshold, olfactory discrimination capacity and odour identification. | 24 months
  Describe the olfactory performance
To characterise the persistence of SARS-CoV-2 in the olfactory epithelium. | 24 months
  Characterisation of the presence of SARS-CoV-2 by PCR in the olfactory mucosa.
To characterise any damage to the olfactory nerve | 24 months
  Mapping analysis of the olfactory nerve of COVID-19 patients by MRI tractography technique.
To identify the presence of inflammatory markers in patients. | 24 months
  Measurement of cellular and inflammatory markers in the olfactory mucosa.
Detection and measurement of markers of neurological disorders in the blood. | 24 months
  To identify the neurological damage in patients.
Measurement of patients' cognitive performance by neuropsychological assessment (standardised tests). | 24 months
  To identify possible cognitive abnormalities in these patients with prolonged loss of smell.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie Lledo, Prof., Study Director — Institut Pasteur
Locations (1):
- Hôpital Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: No